CLINICAL TRIAL: NCT00548119
Title: A Randomized Comparison of NeoCart to Microfracture for the Repair of Articular Cartilage Injuries in the Knee
Brief Title: NeoCart Phase 2 Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Histogenics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6-01
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Articular Cartilage Damage
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeoCart (Experimental)
  Interventions: Biological: NeoCart
- microfracture (Active Comparator)
  Interventions: Procedure: microfracture

INTERVENTIONS:
Biological: NeoCart — autologous tissue implant
  Arms: NeoCart
Procedure: microfracture — microfracture
  Arms: microfracture

SUMMARY:
The objective of this study is to gather additional information regarding the performance of NeoCart to fill articular cartilage defects in the knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptomatic knee pain indicative of an articular cartilage injury and able and willing to give informed consent.

Exclusion Criteria:

* Patients with any previous surgical treatment other than debridement or microfracture of the study cartilage defect.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2009-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The safety and preliminary efficacy of NeoCart will be compared to conventional microfracture therapy. | One year

SECONDARY OUTCOMES:
This study will extend the experience derived from our Phase 1 study. | One year

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSF, San Francisco, California
  - TRIA Orthopedic Center, Bloomington, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Keller Army Community Hospital, West Point, New York
  - Duke Sports Medicine Center, Durham, North Carolina
  - OHSU, Portland, Oregon

REFERENCES:
- [Derived] Anderson DE, Williams RJ 3rd, DeBerardino TM, Taylor DC, Ma CB, Kane MS, Crawford DC. Magnetic Resonance Imaging Characterization and Clinical Outcomes After NeoCart Surgical Therapy as a Primary Reparative Treatment for Knee Cartilage Injuries. Am J Sports Med. 2017 Mar;45(4):875-883. doi: 10.1177/0363546516677255. Epub 2017 Jan 9. PMID 28068480